CLINICAL TRIAL: NCT04664699
Title: Comparison of Standard Monitoring and Plethysmographic Variability Index-Guided Fluid Therapy In Severe Traumatic Brain Injury Patients Scheduled for Emergency Craniotomies: A Randomised Control Trial
Brief Title: Randomized Control Trial to Compare Standard Monitoring and Plethysmographic Variability Index-Guided Fluid Therapy In 64 Severe Traumatic Brain Injury Patients, Aged 18 to 60 Years Old Undergoing Emergency Craniotomies
Acronym: PVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Radha Ramanathan, Dr, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 19010085
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Severe Traumatic Brain Injury
Keywords: Plethysmographic variability index; standard monitoring; emergency craniotomies
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: This is a single centre, with equal randomisation, single blind, parallel group study conducted in Hospital Universiti Sains Malaysia
Who Masked: Care Provider
Masking Description: next of kin were blinded to the allocated arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plethysmographic Variability Index group (Other): 32 patients who presented to emergency department HUSM diagnosed with severe traumatic brain injury who were randomly assigned to the PVI group
  Interventions: Device: Plethymographic Variability Index
- Standard monitoring group (Other): 32 patients who presented to emergency department HUSM diagnosed with severe traumatic brain injury who were randomly assigned to the standard monitoring group
  Interventions: Device: Standard Monitoring

INTERVENTIONS:
Device: Plethymographic Variability Index — All patients were monitored with the electrocardiogram (ECG), Non Invasive Blood Pressure (NIBP), Pulse oximetry (SpO2) and invasively with an arterial line and central venous line as per institutional protocol. In the PVI group, a pulse oximetry probe was connected to the fourth finger of the hand that did not have an arterial cannulation. The pulse oximeter was connected to a monitor The Massimo ® pulse oximeter (Massimo Corp., Irvine, CA, USA), which has a module for PVI measurements.
  PVI ≥13% indicates volume responsiveness, and PVI < 13% indicates adequate volume
  Arms: Plethysmographic Variability Index group
Device: Standard Monitoring — All patients were monitored with the electrocardiogram (ECG), Non Invasive Blood Pressure (NIBP), Pulse oximetry (SpO2) and invasively with an arterial line and central venous line as per institutional protocol. Patients were resuscitated according to mean arterial pressure/ heart rate and urine output.
  Arms: Standard monitoring group

SUMMARY:
This randomized control trial aims to assess if Plethysmographic Variability Index (PVI)-based therapy improves patient outcome in terms of reduced amount and type of fluid used, lower postoperative lactate levels, lesser increment in sodium and chloride levels, improvement of blood gases in term of pH and BE, and reduction in serum creatinine as compared to standard monitoring based therapy in patients with severe traumatic brain injury.

DETAILED DESCRIPTION:
This is a single centre, with equal randomisation, single blind, parallel group study conducted in Hospital Universiti Sains Malaysia. The physician allocated to the standard monitoring or PVI group were aware of the allocated arm, wherelse the next of kin were blinded to the allocated arm.

This study took place in Hospital Universiti Sains Malaysia , Kubang Kerian , Kelantan from July 2019 Until October 2020. Patient who presented to emergency department HUSM diagnosed with severe traumatic brain injury based on a GCS ( Glasgow Coma Scale ≤ 8), Brain CT Scan finding (based on Marshall and Rotterdam scoring), and the SAPS (simplified acute physical injury) score and were planned for craniotomies were assessed for eligibility.

Randomisation sequence was already created using the online randomisation application. (www.randomizer.org), with a 1:1 allocation by the primary investigator. Once a patient with severe traumatic brain injury has been posted for an emergency craniotomy, a white envelope was given to the anesthetic medical officer, If the patient fulfils the eligibility criteria, and the next of kin have consented for recruitment to this study, a second sealed white envelope will be given to the anesthetic medical officer in charge, which contains data collection sheets and protocols. The envelope given was sequentially numbered and sealed , with the patients name, identity card, and date of enrolment written on it by the physician. These sealed white envelopes, with the PVI machine was kept in a locked cupboard in the Anesthesia department in Hospital Universiti Sains Malaysia, only accessible to the primary investigator.

Doctors in charge will be given a separate protocol for PVI based and Standard monitoring based which acts a a guide for fluid management in patients in from induction of anesthesia ( 0 H) and 24 hours post induction in the Intensive Care Unit (ICU) (24 H). Data was then collected by the principle investigator at the end of 24 hours, or reevaluated earlier if any adverse reaction was reported by the doctor in charge.

The sample size calculation was performed using Power and Sample Size Calculations System, . From the study by Tat in 2016, the standard deviation for amount of fluid used was 2637.45, with a mean difference of 1361.31. The α value is set at 0.05 and power of study at 80%. The sample size is calculated using t test. Adding a drop out rate of 10%, the number in each arm will be 34. All statistical analysis was performed using Statistical Package for the Social Science (SPSS) version 26. Results were presented as frequency (percentages) for descriptive data, mean ( standard deviation) for total fluids as well as mean (confidence interval) for laboratory parameters.

A total of 64 patient were deemed eligible. The demographic data in between groups were analyzed using descriptive analysis chi square test. Independent t-test was used to analyze the total volume and different types of fluid used. The difference in lactate, pH, BE, Sodium and Chloride- and Creatinine between groups was analysed using the Independent t-test.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are between 18-60 years old
* ASA (American Society of Anaesthesiology)I and II
* Diagnosed with Severe Traumatic Brain Injury (based on a GCS ( Glasgow Coma Scale ≤ 8) , intubated and consented for neurosurgeries

Exclusion Criteria:

* Patients with serious cardiac arrhythmias
* Patients with peripheral artery disease
* Presence of renal or liver dysfunction
* Presence of concurrent thoracic injury requiring higher ventilator settings with tidal volume > 10 ml/kg or PEEP > 10
* Presence of extracranial major vascular injury ( upper limb, lower limb, intrathoracic or intrabdominal )
* Patients with no valid consent from next of kin or caretaker

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Types and amounts of fluids used | 0 and 24 hours
  To compare the total amount and types of fluids (crystalloid, colloid and blood) used in both groups at induction of anaesthesia until at the end of 24 hours

SECONDARY OUTCOMES:
Blood lactate | 0 and 24 hours
  To compare the mean difference in blood lactate levels in both at induction and at the end of 24 hours
Sodium and chloride | 0 and 24 hours
  To compare serum electrolytes (sodium and chloride) levels of both groups at induction and at the end of 24 hours
pH and base excess | 0 and 24 hours
  To compare pH and base excess of both groups at induction and at the end of 24 hours
Creatinine | 0 and 24 hours
  To compare serum creatinine of both groups at induction and at the end of 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvis-Miranda HR, Castellar-Leones SM, Moscote-Salazar LR. Intravenous Fluid Therapy in Traumatic Brain Injury and Decompressive Craniectomy. Bull Emerg Trauma. 2014 Jan;2(1):3-14. PMID 27162857
- [Background] Pinsky MR, Payen D. Functional hemodynamic monitoring. Crit Care. 2005;9(6):566-72. doi: 10.1186/cc3927. Epub 2005 Nov 22. PMID 16356240
- [Background] Guerin L, Monnet X, Teboul JL. Monitoring volume and fluid responsiveness: from static to dynamic indicators. Best Pract Res Clin Anaesthesiol. 2013 Jun;27(2):177-85. doi: 10.1016/j.bpa.2013.06.002. PMID 24012230
- [Background] Forget P, Lois F, de Kock M. Goal-directed fluid management based on the pulse oximeter-derived pleth variability index reduces lactate levels and improves fluid management. Anesth Analg. 2010 Oct;111(4):910-4. doi: 10.1213/ANE.0b013e3181eb624f. Epub 2010 Aug 12. PMID 20705785
- [Background] Yu Y, Dong J, Xu Z, Shen H, Zheng J. Pleth variability index-directed fluid management in abdominal surgery under combined general and epidural anesthesia. J Clin Monit Comput. 2015 Feb;29(1):47-52. doi: 10.1007/s10877-014-9567-5. Epub 2014 Feb 21. PMID 24557584
- [Background] Demirel I, Bolat E, Altun AY, Ozdemir M, Bestas A. Efficacy of Goal-Directed Fluid Therapy via Pleth Variability Index During Laparoscopic Roux-en-Y Gastric Bypass Surgery in Morbidly Obese Patients. Obes Surg. 2018 Feb;28(2):358-363. doi: 10.1007/s11695-017-2840-1. PMID 28762023
- [Background] Cesur S, Cardakozu T, Kus A, Turkyilmaz N, Yavuz O. Comparison of conventional fluid management with PVI-based goal-directed fluid management in elective colorectal surgery. J Clin Monit Comput. 2019 Apr;33(2):249-257. doi: 10.1007/s10877-018-0163-y. Epub 2018 Jun 14. PMID 29948666
- [Background] Byon HJ, Lim CW, Lee JH, Park YH, Kim HS, Kim CS, Kim JT. Prediction of fluid responsiveness in mechanically ventilated children undergoing neurosurgery. Br J Anaesth. 2013 Apr;110(4):586-91. doi: 10.1093/bja/aes467. Epub 2012 Dec 18. PMID 23250892
- [Background] Fischer MO, Lemoine S, Tavernier B, Bouchakour CE, Colas V, Houard M, Greub W, Daccache G, Hulet C, Compere V, Taing D, Lorne E, Parienti JJ, Hanouz JL; Optimization using the Pleth Variability Index (OPVI) Trial Group. Individualized Fluid Management Using the Pleth Variability Index: A Randomized Clinical Trial. Anesthesiology. 2020 Jul;133(1):31-40. doi: 10.1097/ALN.0000000000003260. PMID 32205547
- [Background] Liu T, Xu C, Wang M, Niu Z, Qi D. Reliability of pleth variability index in predicting preload responsiveness of mechanically ventilated patients under various conditions: a systematic review and meta-analysis. BMC Anesthesiol. 2019 May 8;19(1):67. doi: 10.1186/s12871-019-0744-4. PMID 31068139
- [Background] Biais M, Cottenceau V, Petit L, Masson F, Cochard JF, Sztark F. Impact of norepinephrine on the relationship between pleth variability index and pulse pressure variations in ICU adult patients. Crit Care. 2011 Jul 12;15(4):R168. doi: 10.1186/cc10310. PMID 21749695
- [Background] Fischer MO, Pellissier A, Saplacan V, Gerard JL, Hanouz JL, Fellahi JL. Cephalic versus digital plethysmographic variability index measurement: a comparative pilot study in cardiac surgery patients. J Cardiothorac Vasc Anesth. 2014 Dec;28(6):1510-5. doi: 10.1053/j.jvca.2014.05.003. Epub 2014 Sep 26. PMID 25263772
- [Background] Chu H, Wang Y, Sun Y, Wang G. Accuracy of pleth variability index to predict fluid responsiveness in mechanically ventilated patients: a systematic review and meta-analysis. J Clin Monit Comput. 2016 Jun;30(3):265-74. doi: 10.1007/s10877-015-9742-3. Epub 2015 Aug 5. PMID 26242233
- [Background] Meng L, Yu W, Wang T, Zhang L, Heerdt PM, Gelb AW. Blood Pressure Targets in Perioperative Care. Hypertension. 2018 Oct;72(4):806-817. doi: 10.1161/HYPERTENSIONAHA.118.11688. No abstract available. PMID 30354725
- [Background] Carney N, Totten AM, O'Reilly C, Ullman JS, Hawryluk GW, Bell MJ, Bratton SL, Chesnut R, Harris OA, Kissoon N, Rubiano AM, Shutter L, Tasker RC, Vavilala MS, Wilberger J, Wright DW, Ghajar J. Guidelines for the Management of Severe Traumatic Brain Injury, Fourth Edition. Neurosurgery. 2017 Jan 1;80(1):6-15. doi: 10.1227/NEU.0000000000001432. PMID 27654000